CLINICAL TRIAL: NCT05181046
Title: Non-inferiority of Nanodropper-mediated Microdrops vs. Standard Drops of 0.5% Timolol Maleate in Patients With Open-angle Glaucoma or Ocular Hypertension
Brief Title: Evaluation of Nanodropper-mediated Microdrops vs. Standard Drops of 0.5% Timolol Maleate in Glaucoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanodropper, Inc. (Industry)
Collaborators: Aravind Eye Care System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: nano001
Record Dates: First submitted 2021-12-16; First posted 2022-01-06 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Glaucoma; Glaucoma, Open-Angle; Glaucoma, Primary Open Angle; Glaucoma and Ocular Hypertension; Ocular Hypertension
Keywords: Glaucoma; Eyedrops; Microdrops
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Standard eyedrops of 0.5% timolol maleate (Active Comparator): Participants randomized to this arm will receive one standard drop of 0.5% timolol maleate in each eye.
  Interventions: Other: Original eyedrop bottle/No Nanodropper
- Nanodropper-mediated microdrops of 0.5% timolol maleate (Experimental): Participants randomized to this arm will receive one microdrop of 0.5% timolol maleate in each eye. Microdrops will be dispensed from bottles with installed Nanodropper adaptors.
  Interventions: Device: Nanodropper adaptor

INTERVENTIONS:
Device: Nanodropper adaptor — The Nanodropper adaptor is a sterile medical device that reduces the size of administered eyedrops by coupling to the original bottle.
  Arms: Nanodropper-mediated microdrops of 0.5% timolol maleate
Other: Original eyedrop bottle/No Nanodropper — The original eyedrop bottle dispenses standard eyedrops.
  Arms: Standard eyedrops of 0.5% timolol maleate

SUMMARY:
The purpose of this study is to evaluate the effect of microdrops vs. standard eyedrops of 0.5% timolol maleate in adults with primary open-angle glaucoma or ocular hypertension in terms of intraocular pressure-lowering efficacy and cardiovascular side effects.

DETAILED DESCRIPTION:
This randomized, single-masked, parallel study aims to evaluate the safety and efficacy of microdrops of 0.5% timolol maleate administered with Nanodropper (experimental intervention) compared to standard drops of 0.5% timolol maleate (active comparator) in patients with primary open-angle glaucoma (OAG) or ocular hypertension (OHT) at Aravind Eye Hospital. At the beginning of the test day, baseline (pre-drug) intraocular pressure (IOP), resting heart rate (HR), and resting systolic and diastolic blood pressure (BP) measurements will be collected. Participants will be randomized to receive standard eyedrops or microdrops of 0.5% timolol maleate (one drop per eye), which will be administered by a trained technician at t = 0. IOP, HR, and BP measurements will be repeated by a masked investigator at t = 1, 2, 5, and 8 hours after drug administration.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Recent diagnosis of primary OAG or OHT
* Treatment-naive (not currently using ophthalmic medication)
* Baseline IOP between 21-35 mm Hg
* Corrected Snellen visual acuity of 6/60 or better in each eye

Exclusion Criteria:

* <18 years old
* A recent history (within the past 6 months) of ocular trauma, infection, or uveitis
* Baseline IOP <21 mm Hg or >35 mm Hg
* History of cardiovascular, pulmonary, cerebrovascular, or chronic renal disease
* History of borderline or uncontrolled systemic arterial hypertension
* Use of any systemic α-agonist or β-blocker within 30 days of study commencement
* History of receiving general anesthesia within the previous 30 days
* Pregnant women and nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2021-11-06 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (mm Hg) | 1 hour after drug administration
Intraocular pressure (mm Hg) | 2 hours after drug administration
Intraocular pressure (mm Hg) | 5 hours after drug administration
Intraocular pressure (mm Hg) | 8 hours after drug administration

SECONDARY OUTCOMES:
Resting heart rate (bpm) | 1 hour after drug administration
Resting heart rate (bpm) | 2 hours after drug administration
Resting heart rate (bpm) | 5 hours after drug administration
Resting heart rate (bpm) | 8 hours after drug administration
Resting systolic and diastolic blood pressure (mm Hg) | 1 hour after drug administration
Resting systolic and diastolic blood pressure (mm Hg) | 2 hours after drug administration
Resting systolic and diastolic blood pressure (mm Hg) | 5 hours after drug administration
Resting systolic and diastolic blood pressure (mm Hg) | 8 hours after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Steger, PhD, Study Director — Nanodropper, Inc.
Locations (2):
- India (2):
  - Aravind Eye Hospital, Madurai
  - Aravind Eye Hospital, Puducherry

IPD SHARING:
Plan to Share IPD: No